CLINICAL TRIAL: NCT03550846
Title: Total Indications Ennovate® Non-Interventional Study on Clinical and Radiological Results With Pedicle Screw Fixation
Brief Title: Clinical and Radiological Investigation of a New Spinal Fixateur Interne (Ennovate®)
Acronym: TENNIS
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1639
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Spinal Fusion
Keywords: Spinal Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is planned and conducted to document all patients in the participating Centers, who are treated with the CE-marked product, the Fixateur Ennovate®, regardless of the diagnosis or indication. Data on performance and safety of the product, validated patient based questionnaires (Oswestry Disability Index, ODI) as well as the satisfaction of the patients in general are captured.

DETAILED DESCRIPTION:
The list of spinal treatments is growing, and healthcare authorities today are at times limiting their access due to a lack of evidence of safety and efficiency.

The study enables a quick, but detailed implant documentation, which is of great interest for the current and future users of the internal fixation system targeted in this study. It includes the relevant outcomes to evaluate safety and efficacy of the implant system for various indications in trauma and degenerative disorders.

ELIGIBILITY:
Inclusion Criteria:

- Consent in the documentation of clinical and radiological results

Exclusion Criteria:

- If it is clear that the patient cannot participate in a follow-up examination, he will be excluded from the study documentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Change of Clinical Results from Preoperative Status to Follow-Up at 12 Months | preoperative, 12 months postoperative
  Clinical Results measured by Oswestry Disability Index (ODI). ODI contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel, each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. Each question is scored on a scale of 0 (indicating the least amount of disability) to 5 5 (indicating most severe disability). The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

CONTACTS AND LOCATIONS:
Overall Officials: Carolin Meyer, Dr., Principal Investigator — Klinik für Orthopädie und Unfallchirurgie der Universitätsklinik Köln
Locations (7):
- Germany (7):
  - APEX Spine Wirbelsäulenpraxis, München, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Carolin Meyer, Cologne
  - Klinik und Poliklinik für Neurochirurgie, Göttingen
  - Katholisches Klinikum Koblenz, Koblenz
  - medius Klinik, Nürtingen
  - Praxis für Neurochirurgie am Klinikum, Tuttlingen